CLINICAL TRIAL: NCT00210054
Title: Pilot Single-Dose Intravenous Pharmacokinetic Evaluation of INS37217 Solution in Healthy Volunteers
Brief Title: A Pharmacokinetic Evaluation Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-105
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — denufosol tetrasodium

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217)

SUMMARY:
The purpose of this trial is to characterize the pharmacokinetics of INS37217 following intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

* are nonsmokers or those subjects whom have not smoked within 6 months
* are within 20% of their ideal body weight
* are healthy on the basis of a pre-trial physical examination

Exclusion Criteria:

* history or suspicion of recent alcohol, barbiturate, amphetamine or narcotic abuse or a positive urine drug test at study screening
* history of cardiac arrhythmias, bronchospastic or cardiovascular disease, diabetes mellitus, thyrotoxicosis, Parkinsonism, or drug allergy
* use of concomitant medication other than hormonal contraceptives and multi-vitamins
* donation of blood in the 60 days preceding the screening visit
* have been diagnosed with HIV, hepatitis B or hepatitis C

Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2002-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
detection and characterization of plasma concentrations of INS37217

SECONDARY OUTCOMES:
Pilot study - not specified

CONTACTS AND LOCATIONS:
Overall Officials: Robin Deterding, MD, Principal Investigator